CLINICAL TRIAL: NCT06093087
Title: Internal Fixation Reconstruction With Stent Screw VS Balloon Kyphoplasty in the Treatment of Kummell's Disease: a Double Blinded Randomized Controlled Trial
Brief Title: Randomized Controlled Trial of Internal Fixation Reconstruction With Stent Screw in the Treatment of Kummell's Disease
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LWL_2023
Record Dates: First submitted 2023-10-19; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: BKP; Osteoporotic Vertebral Compression Fracture; Kummell's Disease; Stent-screw-assisted Internal Fixation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAIF (Experimental): patients will be treated with kyphoplasty surgery combined with pedicular screw-assisted internal fixation for vertebral augmentation
  Interventions: Procedure: SAIF
- BKP (Active Comparator): patients will be treated with balloon kyphoplasty surgery for vertebral augmentation
  Interventions: Procedure: BKP

INTERVENTIONS:
Procedure: SAIF — The patient was placed in a prone position under general anesthesia. Using a C-arm X-ray machine and a positioning plate for navigation, the target position on the vertebral body was located one the surface of the body. The puncture needle core was withdrawn after puncturing, and a guide needle was inserted. After removing the puncture needle sleeve, a hollow bone cement screw was screwed into the anterior column of the vertebral body through the guide needle. Subsequently, bone cement was injected into the appropriate position through the bone cement screw to restore the vertebral height
  Arms: SAIF
Procedure: BKP — The patient was placed in a prone position after general anesthesia. Using a C-arm X-ray machine and a positioning plate for guidance, the target position on the vertebral body was located from the surface of the body. A puncture needle sleeve was inserted into the vertebral body. A PKP balloon was then inserted to perform vertebral restoration. After removing the balloon, an appropriate amount of bone cement was injected to ensure even distribution within the vertebral body. Vertebral height augmentation and restoration will then be achieved.
  Arms: BKP

SUMMARY:
This study is a multicenter, prospective, double-blind, randomized controlled trial using a parallel two-arm design to investigate whether the postoperative 6-month quality of life, vertebral stability, complication of patients with osteoporotic vertebral compression fractures (Kummell's disease) are better with the use of stent screw internal fixation and percutaneous bone cement reconstruction technique compared to patients undergoing traditional percutaneous balloon kyphoplasty (BKP) for vertebral augmentation

ELIGIBILITY:
Inclusion Criteria:

* Age 60 or above, gender not specified.
* Must have one to three vertebral segments with vertebral compression fracture (VCF) located between T5 and L5, attributed to underlying primary or secondary osteoporosis rather than cancer.
* All VCFs must exhibit the following radiographic changes: according to Genant's criteria, acute (≤4 months) decrease in anterior, middle, or posterior vertebral height by at least one grade (20-25% reduction in vertebral height, 10-20% reduction in vertebral area) compared to previous X-ray, CT, or MRI results.
* All VCFs for treatment must occur within four months or less.
* All VCFs for treatment must be technically feasible and clinically suitable for BKP or SAIF surgery.
* Pre-treatment back pain NRS score must be ≥ 7 and ineffective with conservative (non-surgical) treatment.
* Pre-treatment Oswestry Disability Index must be ≥ 30 (on a scale of 0-100).
* Patient's life expectancy must be ≥ 12 months.
* Must declare willingness to participate in all post-operative follow-ups.
* Must be capable of understanding the risks and benefits of the study and willing to provide written informed consent.

Exclusion Criteria:

* Vertebral morphology or fracture morphology unsuitable for balloon kyphoplasty. VCF caused by high-energy trauma.
* Asymptomatic VCF or vertebral bodies amenable to prophylactic treatment.
* VCF at the same site associated with primary bone tumors.
* Back pain caused by reasons other than acute fractures. VCF with an estimated fracture time of more than 4 months, based on clinical assessment (radiological evidence and patient history).
* VCF associated with secondary radiculopathy or neurological compromise.
* VCF requiring spinal surgery other than BKP or SAIF.
* Spinal cord compression or vertebral canal injury requiring decompression surgery.
* Combined clinical conditions unsuitable for surgery or affecting subsequent long-term data collection or follow-up.
* Allergy to any component during the surgical procedure (e.g., bone cement, contrast agents).
* Concurrent participation in another clinical study.
* Pregnancy during the study or planning to become pregnant.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
ODI score | ODI score measured 1,3,6 months post surgery during follow up
  Each patients were asked to complete the Oswestry Disability Index questionnaire postoperatively during follow up

SECONDARY OUTCOMES:
CT imaging indicators related to vertebral body stability | all variables were measured 1,3,6 months post surgery during follow up
  There are total 5 indicators measured based on CT images: Anterior vertebral height (ant VBH), middle vertebral height (mid VBH), posterior vertebral height (post VBH), vertebral kyphosis angle (VKA), local kyphosis angle (LKA)
SF36 score | measured 1,3,6 months post surgery during follow up
  SF-36 questionnaire aimed at two different constructs to measure health-related quality of life: the Physical Component and the Mental Component
VAS score | measured 1,3,6 months post surgery during follow up
  The Visual Analogue Scale (VAS) measures pain intensity. 0 indicates no pain and 10 indicates pain as bad as it could possibly be
EQ-5D score | measured 1,3,6 months post surgery during follow up
  The EQ-5D descriptive system measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.